CLINICAL TRIAL: NCT01774045
Title: A Dose Escalation Phase I Study of PDC-1421 Capsule to Evaluate the Safety in Healthy Volunteers
Brief Title: A Dose Escalation Phase I Study of PDC-1421 Capsule Targeting in Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioLite, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Phase I study of PDC-1421
Record Dates: First submitted 2013-01-20; First posted 2013-01-23 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2014-09

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PDC-1421 (Experimental): Dosage form: 380mg PDC-1421 per Capsule. Dosage: single dose (1, 3, 6, 10 capsule(s)). Frequency: once daily, p.o., after meal. Duration: single dose at Day 1, and observing for three Days.
  Interventions: Drug: PDC-1421
- Placebo control (Placebo Comparator): Dosage form: Capsule. Dosage: single dose (1, 3, 6, 10 capsule(s)). Frequency: once daily, p.o., after meal. Duration: single dose at Day 1, and observing for three Days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PDC-1421
  Arms: PDC-1421
Drug: Placebo
  Arms: Placebo control

SUMMARY:
The purpose of this study is to evaluate the safety of PDC-1421 Capsule in healthy subject, find the effective adequate dose for the next stage of the study, and accumulate information of possible mechanism of its anti-depressive effect.

DETAILED DESCRIPTION:
Outcome measures: Physical examination, Vital sign, Electrocardiograph (ECG), Hematology, Blood chemistry, AEs/SAEs monitoring and Columbia-Suicide Severity Rating Scale (C-SSRS)

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-65 years.
2. Subjects must be able to understand and willing to sign informed consent.
3. Female subjects of child-bearing potential must test negative to pregnancy and use appropriate birth control method from the beginning of study to the 15 days later after ending of study.
4. Laboratory data: red blood cell count(RBC),white blood cell count(WBC), platelets, hematocrit, hemoglobin, prothrombin time(PT), partial thromboplastin time (aPTT),aspartate transaminase(AST),alanine aminotransferase(ALT), Lactate dehydrogenase(LDH), total bilirubin, blood urea nitrogen(BUN),serum creatinine, free thyroxine (FT4), thyroid-stimulating hormone (TSH) level,sodium, potassium, calcium, glucose, are all within the normal range.
5. No significantly abnormal findings on physical examination, ECG and vital sign.

Exclusion Criteria:

1. With any clinically significant neurological, gastrointestinal, renal, hepatic,cardiovascular, respiratory, metabolic, endocrine, hematological or other major disorders as determined by the Investigator.
2. A positive drug screen.
3. Any mental disorder diagnosed by board-certificated psychiatrist through detailed diagnostic interview.
4. Any history of suicidal behavior in the past 6 months when evaluated by the C-SSRS.
5. The intensity of suicidal ideation in the past 6 months is no less than 4 defined by the C-SSRS.
6. Have received any prescribed medicine, investigational drug or any non prescribed medicine (including herbal remedies) with 14 days prior to enroll this study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Ta Li, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Tung-Ping Su, M.D, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- PDC-1421: Dosage form: 380mg PDC-1421 per Capsule. Dosage: single dose (1, 3, 6, 10 capsule(s)). Frequency: once daily, p.o., after meal. Duration: single dose at Day 1, and observing for three Days.
  PDC-1421
- Placebo Control: Dosage form: Capsule. Dosage: single dose (1, 3, 6, 10 capsule(s)). Frequency: once daily, p.o., after meal. Duration: single dose at Day 1, and observing for three Days.
  Placebo
Period: Overall Study
Arm/Group | PDC-1421 | Placebo Control
Started | 23 | 7
Completed | 23 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject administrated with 380mg PDC-1421 lost baseline values of hematology and blood chemistry due to hemolysis and the problem never happens again after the nurse corrected her method of drawing blood. We reported this situation to DSMB and they suggested the remaining data to be included in ITT data set and agreed to enroll new subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | PDC-1421 | Placebo Control | Total
Number analyzed (Participants) | 23 | 7 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (3.3) | 27.2 (3.5) | 26.8 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 14 | 6 | 20
Region of Enrollment [Number; unit: participants]
  Taiwan | 23 | 7 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicity of Physical Examination
Description: Physical examination, including skin, head, neck, eyes, ears, nose, throat, heart, lungs, abdomen (liver and spleen), neurological examination, lymph node and extremities, is measured at each visit from screening to follow-up.
Time Frame: baseline to 72 hours
Measure: Number; unit: participants
Groups:
- PDC-1421: Dosage form: 380mg PDC-1421 per Capsule. Dosage: single dose (1, 3, 6, 10 capsule(s)). Frequency: once daily, p.o., after meal. Duration: single dose at Day 1, and observation from baseline to the following 72 hours
- Placebo Control: Dosage form: Capsule. Dosage: single dose (1, 3, 6, 10 capsule(s)). Frequency: once daily, p.o., after meal. Duration: single dose at Day 1, and observation from baseline to the following 72 hours.
Arm/Group | PDC-1421 | Placebo Control
Number analyzed (Participants) | 23 | 7
participants | 0 | 0

2. Primary Outcome: Number of Dose Limiting Toxicity of Electrocardiograph
Description: Electrocardiograph (ECG) is measured at each visit. At visit 2, subjects were measured at 1,2, 4, 8, 12 and 24 hours after drug administration.
Time Frame: baseline to 72 hours
Measure: Number; unit: participants
Groups:
- Placebo Control: Dosage form: Capsule. Dosage: single dose (1, 3, 6, 10 capsule(s)). Frequency: once daily, p.o., after meal. Duration: single dose at Day 1, and and observation from baseline to the following 72 hours
Arm/Group | PDC-1421 | Placebo Control
Number analyzed (Participants) | 23 | 7
participants | 0 | 0

3. Primary Outcome: Number of Dose Limiting Toxicity of Vital Sign
Description: Vital sign, including heart rate, blood pressure and body temperature, are measured at each visit and at 1,2,3,4,8,12 and 24 hours after drug administration.
Time Frame: baseline to 72 hours
Measure: Number; unit: participants
Arm/Group | PDC-1421 | Placebo Control
Number analyzed (Participants) | 23 | 7
participants | 0 | 0

4. Primary Outcome: Number of Dose Limiting Toxicity of Laboratory Values
Description: Laboratory tests are composed of hematology and blood chemistry and measured at each visit. Hematology are composed of RBC, WBC, platelets, hematocrit, hemoglobin, prothrombin time (PT) and partial thromboplastin time (aPTT). Blood chemistry are composed of AST, ALT, LDH, total bilirubin, BUN, serum creatinine, free thyroxine (FT4), TSH, sodium, calcium, potassium, glucose, LDL, HDL, cholesterol and HbA1c.
Time Frame: baseline to 72 hours
Measure: Number; unit: participants
Arm/Group | PDC-1421 | Placebo Control
Number analyzed (Participants) | 23 | 7
participants | 0 | 2

5. Primary Outcome: Number of Dose Limiting Toxicity of Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is composed of suicidal ideation, intensity of ideation and suicidal behavior and measured at each visit.
Time Frame: baseline to 72 hours
Measure: Number; unit: participants
Arm/Group | PDC-1421 | Placebo Control
Number analyzed (Participants) | 23 | 7
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | PDC-1421 | Placebo Control
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/7
Other Adverse Events (participants affected / at risk) | 3/23 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDC-1421 (N=23) | Placebo Control (N=7)
Abdominal fullness (Gastrointestinal disorders) | 2 (2) | 1 (1) — This adverse event is mild and 25-50% related to the study drug by principal investigator's judgement. The subjects were recovered during the trial and without treatment intervention.
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — This adverse event is mild and 50% related to the study drug by principal investigator's judgement. The subject was recovered during the trial and without treatment intervention.
Drowsiness (Nervous system disorders) | 0 (0) | 1 (1) — The adverse event is mild and 25-30% related to the study drug by principal investigator's judgement. The subject was recovered during the trial and without treatment intervention.
Sleepiness (Nervous system disorders) | 1 (1) | 1 (1) — The adverse event is mild and 50% related to the study drug by principal investigator's judgement. The subjects were recovered during the trial and without treatment intervention.
Oral ulcer (Nervous system disorders) | 1 (1) | 0 (0) — The adverse event is mild and 25-30% related to the study drug by principal investigator's judgement. The subject was recovered after one week of the end of trial and without treatment intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No